CLINICAL TRIAL: NCT06573697
Title: Treatment of Electroacupuncture with Different Waveform for Subacute Peripheral Facial Paralysis:study Protocol for a Randomized Controlled Trial
Brief Title: EA Treatment with Different Waveform for Subacute BP:study Protocol for a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jing Sun, Deputy director of the teaching department, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GZY-ZJ-KY-23071
Record Dates: First submitted 2024-08-24; First posted 2024-08-27 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-09

CONDITIONS: Bell Palsy
Keywords: Bell palsy; Peripheral facial paralysis; Clinical study; Acupuncture treatment
MeSH Terms: conditions — Bell Palsy; Facial Paralysis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- low-frequency continuous wave group (Experimental): In each treatment session, the patients will receive EA treatment. The selected acupoints for needling will be BL2, GB1, GB14, ST2, SI18, ST6, ST4, ST7, SJ17, EX-HN16, EX-HN5, on affected side, and LI4, bilaterally. After the de-qi sensation is achieved, electrical stimulator will be connected to BL2-GB1, and ST4-ST6, and 2Hz continuous wave will be used for 20 min.
  Interventions: Other: low-frequency continuous wave EA
- discontinuous wave group (Experimental): In each treatment session, the patientss will receive EA treatment. The selected acupoints for needling will be BL2, GB1, GB14, ST2, SI18, ST6, ST4, ST7, SJ17, EX-HN16, EX-HN5, on affected side, and LI4, bilaterally. After the de-qi sensation is achieved, electrical stimulator will be connected to BL2-GB1, and ST4-ST6, and 40Hz discontinuous wave will be used for 20 min.
  Interventions: Other: discontinuous wave EA
- dilatational wave group (Experimental): In each treatment session, the patientss will receive EA treatment. The selected acupoints for needling will be BL2, GB1, GB14, ST2, SI18, ST6, ST4, ST7, SJ17, EX-HN16, EX-HN5, on affected side, and LI4, bilaterally. After the de-qi sensation is achieved, electrical stimulator will be connected to BL2-GB1, and ST4-ST6, and 2/100Hz dilatational wave will be used for 20 min.
  Interventions: Other: dilatational wave EA

INTERVENTIONS:
Other: low-frequency continuous wave EA — In each treatment session, the subjects will receive EA treatment. The selected acupoints for needling will be BL2, GB1, GB14, ST2, SI18, ST6, ST4, ST7, SJ17, EX-HN16, EX-HN5, on affected side, and LI4, bilaterally. After the de-qi sensation is achieved, electrical stimulator will be connected to BL2-GB1, and ST4-ST6, and 2Hz continuous wave will be used for 20 min.
  Arms: low-frequency continuous wave group
Other: discontinuous wave EA — In each treatment session, the subjects will receive EA treatment. The selected acupoints for needling will be BL2, GB1, GB14, ST2, SI18, ST6, ST4, ST7, SJ17, EX-HN16, EX-HN5, on affected side, and LI4, bilaterally. After the de-qi sensation is achieved, electrical stimulator will be connected to BL2-GB1, and ST4-ST6, and 40Hz discontinuous wave will be used for 20 min.
  Arms: discontinuous wave group
Other: dilatational wave EA — In each treatment session, the subjects will receive EA treatment. The selected acupoints for needling will be BL2, GB1, GB14, ST2, SI18, ST6, ST4, ST7, SJ17, EX-HN16, EX-HN5, on affected side, and LI4, bilaterally. After the de-qi sensation is achieved, electrical stimulator will be connected to BL2-GB1, and ST4-ST6, and 2/100Hz dilatational wave will be used for 20 min.
  Arms: dilatational wave group

SUMMARY:
Bell palsy (BP) is a relatively common clinical disease, which leads to functional and esthetic disturbances for patients and results in a lowered quality of life. Electroacupuncture received attention in the management of BP. The aim of this study is to evaluate the curative effect of different waveform of electroacupuncture on peripheral facial paralysis in subacute stage and to screen out the optimal waveform.

DETAILED DESCRIPTION:
This parallel-group, multicenter randomized clinical trial (RCT) will be conducted at the outpatient clinic of three hospitals in China.A total of seventy-five eligible patients will be randomly divided into low frequency continuous wave(n=25) ,discontinuous wave(n=25) and dilatational wave (n=25) groups.All groups will receive traditional acupuncture treatment at selected acupoints (BL2,GB1,GB14,ST2,SI18,ST4,ST6,ST7,SJ17,EX-HN16,EX-HN5,LI4),additionally,receive different waveform of electroacupuncture treatment for 20 minutes three times per week for four weeks.Facial Nerve Grading System 2.0 (FNGS 2.0) will be used to assess the curative effect at baseline and at 4 weeks after treatment, as the primary outcome.Sunnybrook facialgrad-ingsystem(SFGS) and Facial Disability Index (FDI)Scale will be measured and analyzed at baseline and at 4 weeks after treatment, as secondary outcomes.In addition,amplitude ratio of the affected/healthy side will be another secondary outcome tested by ENoG at bsaeline.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meet the clinical classification criteria for BP, diagnosed by specialist.
2. 1-3 weeks from onset.
3. Male or female patients aged 18-65 years.
4. FNGS2.0≥4
5. Clearly aware, able to complete normal communication, signed informed consent.

Exclusion Criteria:

1. Facial paralysis due to other causes, such as stroke, Guillain-Barre syndrome, multiple sclerosis, encephalitis, facial nerve tumors, skin tumors, parotid tumors, and facial nerve trauma;.
2. Patients with Hunter's syndrome.
3. Patients with bilateral facial nerve palsy.
4. Patients with hemifacial spasm as the the main clinical symptoms.
5. Patients with severe cardiovascular and cerebrovascular diseases, liver, kidney, hematopoietic system diseases, malignant tumors and systemic organ failure, pregnant or lactating patients.
6. Patients with a tendency to bleed easily, who are not suitable for electroacupuncture such as installing a pacemaker, or who cannot cooperate with treatment for other reasons.
7. Participants in other clinical trials within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline score of the Facial Nerve Grading System 2.0(FNGS 2.0) | Baseline,4 weeks
  Evaluation of the facial nerve function using the Facial Nerve Grading System 2.0 (FNGS 2.0). In the FNGS 2.0, the minimal score is 4, which indicates normal function, and the maximal score is 24, which indicates the worst function.

SECONDARY OUTCOMES:
Change from Baseline score of the Sunnybrook grading(SFGS) scale | Baseline,4 weeks
  The Sunnybrook grading scale includes 3 subscales, which are the resting symmetry subscale, the symmetry of voluntary movement subscale, and the synkinesis subscale. In the resting symmetry subscale, the minimal score is 0, which indicates normal resting symmetry, and the maximal score is 20, which indicates the most severe resting asymmetry. In the symmetry of voluntary movement subscale, the minimal score is 20, which indicates gross asymmetry of voluntary movement, and the maximal score is 100, which indicates normal symmetry of voluntary movement. And in the synkinesis subscale, the minimal score is 0, which indicates no involuntary muscle contraction associated with each expression, and the maximal score is 15, which indicates the most severe involuntary muscle contraction associated with each expression. The composite score equals to the symmetry of voluntary movement score minus the resting symmetry score and the synkinesis score.
Change from Baseline score of the Facial Disability Index(FDI) | Baseline,4 weeks
  The FDI is a brief, self-report questionnaire of physical disability and psychosocial factors related to facial neuromuscular function. It was intended to assess disability and the outcome of intervention in terms of meaningful change in the patient's physical disability and psychosocial status.
Change from Baseline value of the amplitude ratio of the compound muscle action potential (CMAP) of the affected side in the ENoG test. | Baseline
  Change from Baseline value of the amplitude ratio of the compound muscle action potential (CMAP) of the affected side in the ENoG test.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Sun, Ph.D, Principal Investigator — The Third Clinical College of Zhejiang Chinese Medical University
Locations (1):
- The Third Affiliated hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No